CLINICAL TRIAL: NCT05765396
Title: SARS-CoV-2/COVID-19 Study of Next Generation Non-Invasive Passive Detection Technologies
Acronym: PassiveDetect
Status: Active, not recruiting | Type: Observational
Sponsor: The Geneva Foundation (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency); Level 42 AI, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C.2023.007
Record Dates: First submitted 2023-03-09; First posted 2023-03-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-08

CONDITIONS: COVID-19; SARS-CoV-2 Virus; COVID-19 Pneumonia; COVID-19 Respiratory Infection; COVID-19 Acute Respiratory Distress Syndrome; Corona Virus Infection; Influenza; RSV Infection
Keywords: COVID-19 diagnostic product, e-stethoscope, military, Flu, RSV, Passive Detection, Level 42
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Influenza, Human; Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19, Flu, and/or RSV positive patients: Participants screened with known COVID-19, Flu, and/or RSV positive test results obtained within 48hrs of recruitment.
  Interventions: Device: imPulse™ Systems (Una and TOR) infrasound-to-ultrasound e-stethoscope
- COVID-19, Flu, and/or RSV negative patients: Participants screened with known COVID-19, Flu, and/or RSV negative test results obtained within 48hrs of recruitment.
  Interventions: Device: imPulse™ Systems (Una and TOR) infrasound-to-ultrasound e-stethoscope

INTERVENTIONS:
Device: imPulse™ Systems (Una and TOR) infrasound-to-ultrasound e-stethoscope — The imPulse™ Systems are an every/anywhere-point-of-care cardiopulmonary functional state assessment platform designed to capture normal and abnormal, audible and inaudible cardiopulmonary sounds, rhythms and patterns, via a real-time, intelligent, full-spectrum phonocardiogram obtained from direct to skin coupling or through a layer of clothing.
  Other Names: imPulse™ Una; e-stethoscope; Passive Detection; imPulse™ TOR

SUMMARY:
The goal of this observational study is to evaluate new non-invasive passive surveillance technologies, Level 42 AI imPulse™ Una and TOR devices for the detection of COVID-19, Flu, and/or RSV in asymptomatic and symptomatic individuals over age of 18 undergoing COVID-19, Flu, and/or RSV screening and testing at BAMC Ft Sam Houston, TX; with and without COVID-19, Flu, and/or RSV.

The hypotheses are:

(H1) The imPulseTM Una and the imPulseTM TOR e-stethoscopes have at least a similar discriminative and detection ability among symptomatic and asymptomatic COVID-19 carrier versus those not infected compared to gold standard RT-PCR. We will operationalize and deploy both the imPulseTM Una and imPulseTM TOR e-stethoscope into DoD use-cases and compare their usability between the devices.

(H2) Identify if the imPulseTM Una and the imPulseTM TOR e-stethoscopes have at least a similar discriminative and detection ability among symptomatic and asymptomatic Respiratory Syncytial Virus (RSV), Influenza and Long COVID carriers versus those not infected compared to gold standard Rapid RSV and Flu Antigen Tests, or RT-PCR and molecular assays. We will operationalize and deploy both the imPulseTM Una and imPulseTM TOR e-stethoscope into DoD use-cases and compare their captured traces in the early identification of disease/illness analyzed by the devices built in algorithms.

(H3) In the mid to long-term, this approach will also be explored as a diagnostic system to explore pursue the physical (structural and mechanical) properties of cells and tissues that maintain normal cell behavior (motility, growth, apoptosis), and the critical importance of the ability of cells to sense and respond to mechanical stresses, which will be operationally critical for assessment of both traumatic and unconventional exposures in austere environments.

Participants will:

* Be consented;
* Be screened for COVID-19, Flu, and/or RSV symptoms according to BAMC's current screening procedures;
* Have study data collected;
* Complete a symptoms questionnaire;
* imPulseTM Una and TOR e-stethoscopes examination will be conducted;
* Participants will be compensated for completing all study requirements. (Active-Duty personnel must complete the study procedures while off-duty in order to receive compensation.)

DETAILED DESCRIPTION:
Emerging acute respiratory diseases (ARDs) pose a significant threat for the US military, especially among those in training environments where crowded living conditions and demanding multi-factorial stresses exacerbate infection exposure and suppress immunity, respectively. Consequently, ARD rates are routinely reported higher in recruits than older military personnel, which have a detrimental effect on operational readiness. Although significant steps, such as surveillance and vaccine programs, have been taken to minimize the impact that ARDs have on military recruits and newly mobilized troops, hospitalizations among recruits still exceeds that of comparable civilian population in the United States by at least 3- to 4- folds, accounting for almost 30% of all infectious disease associated hospitalizations. In 2018, respiratory infections like respiratory syncytial virus (RSV), accounted for an estimated 50,000 medical encounters affecting about ~35,000 recruits that resulted in 1,000 hospital bed days leading to significant loss in training time and cost. In addition to annual respiratory infections such as influenza, on-going COVID-19, which has claimed the lives of 210,000 Americans, continues to threaten to further degrade operational readiness. Thus, inexpensive, rapid, and more reliable diagnostics are continually required to better treat and prevent ARDs to preserve military readiness and decrease disability adjusted life years.

Regaining American technological supremacy will require a pivot from the large, exquisite, hardware- defined systems that won us the conflicts of last century to larger numbers of lower-cost, attritable,smaller, software-defined systems. This is particularly critical as the country reopens, and life returns to normal, thus long-term technological technology platforms must be able to secure entry to workplaces, airplanes, schools, stadiums, theaters, mass transit center, ports-of-entry, malls and restaurants.

Current CLIA laboratory diagnostic procedures, such Enzyme Linked Immunosorbent Assay (ELISA), Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), and bacterial cultures, are costly, time- consuming, and operator sensitive. It has become apparent that during the dynamic COVID-19 pandemic, these approaches are insufficient in meeting diagnostic needs as they are difficult to scale-up and lack logistical flexibility. Furthermore, due to the invasive nature of active clinical sampling, there is a critical need for accurate and rapid passive surveillance as to screen for SARS-CoV-19 as well as other hazardous chemical and biological agents. To address this capability gap, the current project will- modify and operationalize existing innovative passive surveillance systems that can be deployed in the near-term.

The Level 42 AI imPulseTM UNA and TOR are both over-clothing e-stethoscope and stand-off systems which are intended to be used to identify characteristic and subtle changes in audible and inaudible sounds changes in the upper and lower respiratory tract driven by airflow velocity, hydration, pressure, and wall shear stress for both inspiration (velocity splitting) and expiration (velocity merging) during active infection vs. health. The Level 42 AI imPulseTM TOR improves upon the UNA and adds the capabiliy to perform non-contact, alternating multi-lead electrocardiogram (ECG) and electromyography (EMG) sensors along with existing broad-spectrum vibroacoustic biosignature sensors. This allows the TOR to collect six types of inaudible vibrations and audible sounds as i) Korotkoff sounds and murmurs, ii) heartbeat, iii) respiratory rhythm, iv) gut motility, v) carotid tree blood flow and resistance, and vi) Traube-Hering waves, which measure states of stress tension.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic and symptomatic individuals 18 years and older
* Receiving standard COVID-19, Flu, and/or RSV screening and testing at BAMC
* Do not have to be diagnosed with SARS-CoV-19 (COVID-19), Flu, and/or RSV but only be screened
* English Speaking

Exclusion Criteria:

* Any individual under age of 18
* Anyone unable to comply (or be assisted) with study procedures
* Anyone not able to provide temperature thermal scan, and/or 3-minute vibroacoustic scan

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asymptomatic and symptomatic individuals age 18 and older undergoing COVID-19, Flu, and/or RSV screening and testing at Brooke Army Medical Center (BAMC), Ft Sam Houston TX, with and without COVID-19, Flu, and/or RSV diagnosis within 48hrs of consent.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Digital vibroacoustic biomarker diagnostic performance characteristics specific to imPulse™ Una | Enrollment through to study completion (min 48hrs through to 24 months)
  Sensitivity, specificity, positive and negative predictive values - of the imPulse™ Una device for point-of-care diagnosis of COVID-19 among symptomatic and asymptomatic COVID-19 carrier versus those not infected compared to gold standard RT-PCR.
imPulse™ Una infrasound-to-ultrasound e-stethoscope device usability | Enrollment through to study completion (min 48hrs through to 24 months)
  Critical importance of the ability to sense and respond to mechanical stresses, which will be operationally critical for assessment of both traumatic and unconventional exposures in austere environments
imPulse™ TOR infrasound-to-ultrasound e-stethoscope device usability | Enrollment through to study completion (min 48hrs through to 24 months)
  Critical importance of the ability to sense and respond to mechanical stresses, which will be operationally critical for assessment of both traumatic and unconventional exposures in austere environments
Digital vibroacoustic biomarker diagnostic performance characteristics specific to imPulse™ TOR | Enrollment through to study completion (min 48hrs through to 24 months)
  Sensitivity, specificity, positive and negative predictive values - of the imPulse™ TOR device for point-of-care diagnosis of COVID-19, Flu, and/or RSV among symptomatic and asymptomatic COVID-19, Flu, and/or RSV carrier versus those not infected compared to gold standard RT-PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Tony T Yuan, PhD, Principal Investigator — Uniformed Services University of the Health Sciences (USUHS); Michael Morris, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clemmons NS, McCormic ZD, Gaydos JC, Hawksworth AW, Jordan NN. Acute Respiratory Disease in US Army Trainees 3 Years after Reintroduction of Adenovirus Vaccine 1. Emerg Infect Dis. 2017 Jan;23(1):95-98. doi: 10.3201/eid2301.161297. Epub 2017 Jan 15. PMID 27748651
- [Background] Sanchez JL, Cooper MJ, Myers CA, Cummings JF, Vest KG, Russell KL, Sanchez JL, Hiser MJ, Gaydos CA. Respiratory Infections in the U.S. Military: Recent Experience and Control. Clin Microbiol Rev. 2015 Jul;28(3):743-800. doi: 10.1128/CMR.00039-14. PMID 26085551
- [Background] Armed Forces Health Surveillance Center (AFHSC). Surveillance Snapshot: illness and injury burdens among U.S. military recruit trainees, 2012. MSMR. 2013 Apr;20(4):24. No abstract available. PMID 23617314
- [Background] Murray CJ, Lopez AD. Measuring the global burden of disease. N Engl J Med. 2013 Aug 1;369(5):448-57. doi: 10.1056/NEJMra1201534. No abstract available. PMID 23902484
- [Background] Alahi MEE, Mukhopadhyay SC. Detection Methodologies for Pathogen and Toxins: A Review. Sensors (Basel). 2017 Aug 16;17(8):1885. doi: 10.3390/s17081885. PMID 28813028